CLINICAL TRIAL: NCT02565472
Title: Effect of a White Grape Juice Compared to Apple Juice on Gastrointestinal Tolerance and Breath Hydrogen Response in Human Subjects
Brief Title: Effects of Juice on Gastrointestinal Tolerance and Breath Hydrogen Response in Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1508M77407
Record Dates: First submitted 2015-09-22; First posted 2015-10-01 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Apple Juice (Experimental): 12 oz apple juice
  Interventions: Other: Apple juice
- Grape Juice (Experimental): 12 oz grape juice
  Interventions: Other: White grape juice

INTERVENTIONS:
Other: White grape juice
  Arms: Grape Juice
Other: Apple juice
  Arms: Apple Juice

SUMMARY:
The goal of this study is to determine subjective gastrointestinal tolerance response and differences in breath hydrogen response following the consumption of two types of juice. This double-blind crossover study requires participants to arrive to the lab 12 hours fasted, consume 12 oz of juice and complete gastrointestinal tolerance questionnaires as well as produce samples for breath hydrogen analysis at various time points over the next 3 hours. Subjects will be asked to complete additional questionnaires at 12 and 24 hours post consumption, from home. Subjects will also be asked to keep a food record for 24 hours prior to their scheduled visit times to assure compliance.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 Body mass index between 18-29 kg/m2 Demonstrates spoken and written English literacy and able to provide written, informed consent after review of study protocol and procedures

Exclusion Criteria:

* • Use of enemas, laxatives, proton pump inhibitors, or antibiotics within the past 3 months

  * Smoker
  * Not a regular breakfast or eater
  * Self-reported history of a past or current gastrointestinal disease
  * High fiber eater (≥3 servings of high fiber foods per day)
  * Concurrent or recent (within 30 days) participation in an intervention trial
  * Recent weight fluctuations
  * Allergies to any of the test products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal tolerance from baseline | 24 hours
  Subjects will answer a 7 symptom questionnaire regarding the intensity of gastrointestinal symptoms experienced following juice consumption. Questionnaire is adapted from the validated Bovenschen gastrointestinal tolerance questionnaire. Questionnaire is to be completed at the following time points: baseline, 30 min, 60 min, 90 min, 120 min, 180 min, 12 hours, 24 hours.

SECONDARY OUTCOMES:
Change in Breath Hydrogen from baseline | 2 hours
  Patients will be asked to exhale a full breath into a sample collection bag. The breath samples will be extracted and measured using the Quintron BreathTracker Analyzer at time points: baseline, 60 min, 120 min. This will be a marker of carbohydrate fermentation in the colon.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States